CLINICAL TRIAL: NCT00622986
Title: A Multicentered RCT Study of the Efficacy and Safety of an Extract of Cimicifuga Foetida L. for the Treatment of Climacteric Symptoms of Chinese Women
Brief Title: China Cimicifuga Trial of Climacteric Complaint Control
Acronym: CCCCC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Luye Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Prof. Lin Shouqing, Beijing Union Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XMT-5Cs-002-2007
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: Climacteric Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1 (Experimental): perimenopausal women
  Interventions: Drug: an extract of Cimicifuga Foetida L.
- A2 (Placebo Comparator): perimenopausal women
  Interventions: Drug: placebo
- B1 (Experimental): early staged postmenopausal women
  Interventions: Drug: an extract of Cimicifuga Foetida L.
- B2 (Placebo Comparator): early staged postmenopausal women
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: an extract of Cimicifuga Foetida L. — Each patient will be given the medication of extract of Cimicifuga Foetida L. 2 tablets each day for 3 months.
  Other Names: Ximingting
  Arms: B1
Drug: an extract of Cimicifuga Foetida L. — Each patient will be given the medication of extract of Cimicifuga Foetida L. 2 tablets each day for 3 months.
  Other Names: Ximingting
  Arms: A1
Drug: placebo — Each patient will be given placebo of 2 tablets each day for 3 months.
  Arms: A2
Drug: placebo — Each patient will be given placebo of 2 tablets each day for 3 months.
  Arms: B2

SUMMARY:
This study is designed to determine whether an extract of Cimicifuga Foetida L. is safe and efficacious to relieve the climacteric symptoms of Chinese women

DETAILED DESCRIPTION:
Extracts of Cimicifuga Racemosa (black cohosh) have been widely used in North America and Europe for decades for the treatment of menopause related problems, either as nutritional supplements or as pharmaceutical products. Previous clinical trials had shown that an extract of Cimicifuga Foetida L.(Ximingting, Luyepharm), which was standardized to have similar components of an extract of Cimicifuga Racemosa, was safe and efficacious to relieve the climacteric symptoms and signs in Chinese women who were recruited according to criteria categorized by theory of Traditional Chinese Medicine.We are interested to know whether it may have the same efficacy and safety profiles when judged with method and standard commonly accepted in western medicine.

ELIGIBILITY:
Inclusion Criteria:

* Having climacteric symptoms with hot flushes >= 3 time per day
* Score of Kupperman Index at baseline >= 20
* In addition to these criteria, women who had menopause longer than 2 months but less than 12 months, with FSH > 15U/L were enrolled into the perimenopausal group. Women having menopause longer than 12 months but less than 5 years, with FSH >= 40U/L and E2 <= 30pg/ml, were assigned into early staged postmenopausal group.

Exclusion Criteria:

* Having history of hysterectomy
* Having HRT within 6 weeks
* Having other drugs or nutritional supplements of relieving climacteric symptoms within one week
* Having psychological counseling within one week
* Having medical history of estrogen-dependent tumors
* The result of pap smear exam at stage III and above
* Having an uterine leiomyoma lager than 4 cm
* The endometrial thickness lager than 0.5 cm
* Having abnormal cardiac, liver or kidney functions
* Having abnormal thyroid function
* Having hypertension, diabetes and coronary heart diseases that were not under control
* Pregnant or suspected pregnant woman
* Having severe mental disorders that inhibit to understand the research purpose
* Other conditions the investigators believed not suitable for enrollment

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Change of scores of Kupperman Index before and after the treatment | 3 months

SECONDARY OUTCOMES:
Change of scores of Menopause Rating Scale before and after the treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shouqing Lin, MD, Study Chair — Beijing Union Hospital
Locations (13):
- China (13):
  - Fujian Provincal Maternal and Children Health Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital，SUN YAT-SEN University, Guangzhou, Guangdong
  - Zhongnan University Xiangya No.3. Hospital, Changsha, Hunan
  - Zhongnan University Xiangya No.2. Hospital, Changsha, Hunnan
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Medical School Hospital Of Qingdao University, Qingdao, Shandong
  - Bejing Union Hospital, Beijing
  - The Great Wall Hospital, Beijing
  - Southwest Hospital, Chongqing
  - Daping Hospital, Chongqing
  - Obstetrics & Gynecology Hospital Of Fudan University, Shanghai
  - International Peace Maternity & Child Health Hospital Of The China Welfare Institute, Shanghai
  - Tianjin City Hospital for Gynaecology and Obsterics, Tianjin